CLINICAL TRIAL: NCT03785314
Title: Effect of Different Posture on Optic Nerve Sheath Diameter During Thoracic Epidural Catheterization
Brief Title: Optic Nerve Sheath Diameter Difference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-11-039
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2019-08

CONDITIONS: Optic Neve Sheath Diameter
Keywords: Optic Nerve Sheath Diameter Different Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection under sitting position (Active Comparator): saline injection under sitting position during thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization
- injection under lateral decubitus position (Active Comparator): saline injection under lateral decubitus position during thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization

INTERVENTIONS:
Other: thoracic epidural catheterization — thoracic epidural catheterization with different posture

SUMMARY:
Intracranial pressure is measured indirectly using optic nerve sheath diameter with ultrasound. It is reported that epidural pressure varies according to different posture ( lateral decubitus vs. sitting position).

This study is designed to measure the optic nerve sheath diameter in lateral decubitus and sitting position, respectively.

DETAILED DESCRIPTION:
According to previous study, injection of different volume of local anesthetics (1.0 ml/kg vs. 1.5 ml/kg) during caudal anesthesia, high volume of local anesthetics resulted in significant increase of intracranial pressure (ICP). Increase of ICP can reduce regional cerebral flow and oxygen saturation causing the safety of patients. In addition, increase of ICP can result in headache, syncope, and transient loss of visual acuity. Although it is very invasive method, ICP can be measured directly at the brain parenchyme. Among methods to measure the ICP indirectly, measurement of optic nerve sheath diameter using ultrasound is known to reflect the degree of ICP. It is reported that optic nerve sheath diameter increases when higher volume of medication is injected during epidural anesthesia. Previous reports showed that epidural pressure varies according to different posture. When epidural pressure was measured in patients of spinal stenosis, lumbar flexion showed lower epidural pressure than epidural pressure of lumbar extension. In addition, when epidural pressure was measured in the sitting position, it showed lower pressure than pressure of lateral decubitus.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level
* previous brain surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter change among 4 time period | Baseline, 10 minutes, 20 minutes, 40 minutes after the completion of the intervention
  optic nerve sheath diameter change among 4 time period using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No